CLINICAL TRIAL: NCT00484718
Title: MEASURES OF GAIT AND SELF-REPORTED PAIN IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE: A RANDOMIZED, SINGLE-BLIND WASHOUT, DOUBLE-BLIND TREATMENT, DOUBLE DUMMY CROSS-OVER PILOT TRIAL USING PLACEBO, OXYCODONE AND CELECOXIB (A9011030)
Brief Title: Measuring Gait And Self-Reported Pain In Patients With Osteoarthritis Of The Knee Using Placebo/Oxycodone/Celecoxib.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A9011030
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: celecoxib
- B (Active Comparator)
  Interventions: Drug: Oxycodone
- C (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celecoxib — oral, 100 mg bid
  Arms: A
Drug: Oxycodone — oral, 20 mg bid
  Arms: B
Drug: placebo — oral bid
  Arms: C

SUMMARY:
The Purpose of this trial is to evaluate the use of a cross-over trial design in an osteoarthritis population. We will determine the inter- and intra-subject variability in osteoarthritis (OA) endpoints and evaluate if efficacy can be detected by measuring OA endpoints following treatment with 2 different types of analgesics in a crossover study of this design.

DETAILED DESCRIPTION:
Methodology study to evaluate the use of a cross over design and gait analysis. The study was terminated by mutual consent with the study site at a meeting on the 1 April 2009, because of slow recruitment due to a high screen fail rate. The study was not stopped for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been taking an NSAID at least 15 of the past 30 days for index knee pain
* Grades 2 or 3 OA as defined by the Kellgren and Lawrence Grading System of the medial tibiofemoral joint (joint space narrowing in the medial compartment > lateral compartment as assessed by x-ray) using the Altman Atlas of OA7. This must be documented with a report from an x-ray of the study joint taken either at screening or within 1 year prior to screening
* Subject meets American College of Rheumatology (ACR) clinical classification criteria for osteoarthritis of the knee, defined by the following: Knee pain and at least 3 of the following: oAge >50 oMorning stiffness <30 minutes oCrepitus on active motion oBony tenderness oBony enlargement oNo palpable warmth of synovium.

Exclusion Criteria:

* Subject has a documented history of an allergic reaction (hives, rash, etc.) or a clinically significant intolerance to celecoxib, sulfonamides, aspirin, or opioids including oxycodone
* Significant pain outside the index knee, including significant hip or back pain that can not be distinguished from OA pain or that interferes with ability to walk. (Patients with bilateral knee OA will be allowed into the study. The index knee should be defined as the more painful knee
* Predominantly patellofemoral knee osteoarthritis in the index knee as assessed by clinical examination
* Subject who are unable to discontinue all formulations of prior analgesics other than acetaminophen during the Washout Period of the study, or who are anticipated to be unable to discontinue rescue medication for 24 hours prior to the respective visits. (Low dose aspirin may be taken for cardiac prophylaxis
* Excessive signal knee joint laxity indicative of functional ligamentous deficiency

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01-17 (Actual); Primary Completion 2009-06-10 (Actual); Study Completion 2009-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - VAPAHCS, Palo Alto, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Asay JL, Boyer KA, Andriacchi TP. Repeatability of gait analysis for measuring knee osteoarthritis pain in patients with severe chronic pain. J Orthop Res. 2013 Jul;31(7):1007-12. doi: 10.1002/jor.22228. Epub 2013 Mar 18. PMID 23508626
- [Derived] Boyer KA, Angst MS, Asay J, Giori NJ, Andriacchi TP. Sensitivity of gait parameters to the effects of anti-inflammatory and opioid treatments in knee osteoarthritis patients. J Orthop Res. 2012 Jul;30(7):1118-24. doi: 10.1002/jor.22037. Epub 2011 Dec 16. PMID 22179861
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011030&StudyName=Measuring%20Gait%20And%20Self-Reported%20Pain%20In%20Patients%20With%20Osteoarthritis%20Of%20The%20Knee%20Using%20Placebo/Oxycodone/Celecoxib.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 6 participants were randomized to receive 1 of 6 possible treatment sequences of ABC, ACB. BAC, BCA, CAB, CBA (where: A=placebo, B=celecoxib, C=oxycodone) in treatment periods 1, 2 and 3 (each 2-week treatment period was separated by a 2-week washout period).
Groups:
- Placebo Then Celecoxib Then Oxycodone: Participants received placebo capsules matched to celecoxib and oxycodone orally, twice daily from Days 1 to 14 of treatment period 1 (participants received placebo from Days 1 to 84 in 3 treatment periods [14 days prior to each treatment periods {i.e. during 2-week washout period}, and Day 1-14 in each treatment period]), then in treatment period 2 participants received celecoxib 100 milligram (mg) (200 milligram per day [mg/day]) capsule orally, twice daily on Days 1-14 followed by oxycodone controlled release 10 mg (20 mg/day) capsule orally, twice daily on Days 1-14 in treatment period 3. Each 2-week treatment period was separated by a 2-week washout period.
- Placebo Then Oxycodone Then Celecoxib: Participants received placebo capsules matched to celecoxib and oxycodone orally, twice daily from Days 1 to 14 of treatment period 1 (participants received placebo from Days 1 to 84 in 3 treatment periods [14 days prior to each treatment periods {i.e. during 2-week washout period}, and Day 1-14 in each treatment period]), then in treatment period 2 participants received oxycodone controlled release 10 mg (20 mg/day) capsule orally twice daily on Days 1-14 followed by celecoxib 100 mg (200 mg/day) capsule orally, twice daily on Days 1-14 in treatment period 3. Each 2-week treatment period was separated by a 2-week washout period.
- Celecoxib Then Placebo Then Oxycodone: Participants received celecoxib 100 mg (200 mg/day) capsule orally, twice daily on Days 1-14 of treatment period 1 then, in treatment period 2 participants received placebo capsules matched to celecoxib and oxycodone orally, twice daily from Day 1 to 14 (participants received placebo from Days 1 to 84 in 3 treatment periods [14 days prior to each treatment periods {i.e. during 2-week washout period}, and Day 1-14 in each treatment period]), followed by oxycodone controlled release 10 mg (20 mg/day) capsule orally, twice daily on Days 1-14 in treatment period 3. Each 2-week treatment period was separated by a 2-week washout period.
- Celecoxib Then Oxycodone Then Placebo: Participants received celecoxib 100 mg (200 mg/day) capsule orally, twice daily on Days 1-14 of treatment period 1, then in treatment period 2 participants received oxycodone controlled release 10 mg (20 mg/day) capsule orally, twice daily on Days 1-14, followed by placebo capsules matched to celecoxib and oxycodone orally, twice daily from Day 1 to 14 of treatment period 3 (participants received placebo from Days 1 to 84 in 3 treatment periods [14 days prior to each treatment periods {i.e. during 2-week washout period}, and Day 1-14 in each treatment period]). Each 2-week treatment period was separated by a 2-week washout period.
- Oxycodone Then Placebo Then Celecoxib: Participants received oxycodone controlled release 10 mg (20 mg/day) capsule orally, twice daily on Days 1-14 in treatment period 1 then, in treatment period 2 participants received placebo capsules matched to celecoxib and oxycodone orally, twice daily from Day 1 to 14 (participants received placebo from Days 1 to 84 in 3 treatment periods [14 days prior to each treatment periods {i.e. during 2-week washout period}, and Day 1-14 in each treatment period]), followed by celecoxib 100 mg (200 mg/day) capsule orally, twice daily on Days 1-14 in treatment period 3. Each 2-week treatment period was separated by a 2-week washout period.
- Oxycodone Then Celecoxib Then Placebo: Participants received oxycodone controlled release 10 mg (20 mg/day) capsule orally, twice daily on Days 1-14 in treatment period 1 then, in treatment period 2 participants received celecoxib 100 mg (200 mg/day) capsule orally, twice daily on Days 1-14, followed by placebo capsules matched to celecoxib and oxycodone orally, twice daily from Day 1 to 14 of treatment period 3 (participants received placebo from Days 1 to 84 in 3 treatment periods [14 days prior to each treatment periods {i.e. during 2-week washout period}, and Day 1-14 in each treatment period]). Each 2-week treatment period was separated by a 2-week washout period.
Period: Treatment Period 1 (2 Weeks)
Arm/Group | Placebo Then Celecoxib Then Oxycodone | Placebo Then Oxycodone Then Celecoxib | Celecoxib Then Placebo Then Oxycodone | Celecoxib Then Oxycodone Then Placebo | Oxycodone Then Placebo Then Celecoxib | Oxycodone Then Celecoxib Then Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Placebo Then Celecoxib Then Oxycodone | Placebo Then Oxycodone Then Celecoxib | Celecoxib Then Placebo Then Oxycodone | Celecoxib Then Oxycodone Then Placebo | Oxycodone Then Placebo Then Celecoxib | Oxycodone Then Celecoxib Then Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (2 Weeks)
Arm/Group | Placebo Then Celecoxib Then Oxycodone | Placebo Then Oxycodone Then Celecoxib | Celecoxib Then Placebo Then Oxycodone | Celecoxib Then Oxycodone Then Placebo | Oxycodone Then Placebo Then Celecoxib | Oxycodone Then Celecoxib Then Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Placebo Then Celecoxib Then Oxycodone | Placebo Then Oxycodone Then Celecoxib | Celecoxib Then Placebo Then Oxycodone | Celecoxib Then Oxycodone Then Placebo | Oxycodone Then Placebo Then Celecoxib | Oxycodone Then Celecoxib Then Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (2 Weeks)
Arm/Group | Placebo Then Celecoxib Then Oxycodone | Placebo Then Oxycodone Then Celecoxib | Celecoxib Then Placebo Then Oxycodone | Celecoxib Then Oxycodone Then Placebo | Oxycodone Then Placebo Then Celecoxib | Oxycodone Then Celecoxib Then Placebo
Started | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants who received at least 1 dose of study medication.
Groups:
- All Participants: All randomized participants who received placebo matched to celecoxib and oxycodone, celecoxib 100 mg and oxycodone 20 mg orally, twice daily in one of the 6 treatment sequences in each of three treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Knee Pain Intensity Measured by Numeric Rating Scale (NRS) at Week 12
Description: The severity of arthritis pain in participant's signal knee at the time of the visit was assessed using an 11-point NRS, ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate worse pain.
Time Frame: Baseline, Week 12
Population: As study was terminated, data for this outcome measure was not collected and analyzed due to low number of participant enrolled which were required to carry out the pre-specified efficacy analysis.
Groups:
- Placebo: Participants received placebo capsules matched to celecoxib and oxycodone orally, twice daily from Day 1 to 84 (Days 1-14 of treatment periods 1, 2, 3 and for 14 days prior to each of three treatment periods [i.e. during 2-week washout period])
- Celecoxib 100 mg: Participants received celecoxib 100 mg (200 mg/day) capsule orally, twice daily on Days 1-14 in each of three treatment periods (each 2-week treatment period was separated by a 2-week washout period).
- Oxycodone 20 mg: Participants received oxycodone controlled release 10 mg (20 mg/day) capsule orally, twice daily on Days 1-14 in each of three treatment periods (each 2-week treatment period was separated by a 2-week washout period).
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Knee Pain Intensity Measured by Visual Analog Scale (VAS) at Week 12
Description: The severity of arthritis pain in participant's signal knee was assessed using a 100-millimeter (mm) VAS ranging from 0 mm = no pain and 100 mm = most severe pain. Higher score indicate more pain.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Change From Baseline in Western Ontario and McMaster (WOMAC) Osteoarthritis Index Pain Subscale Score at Week 12
Description: WOMAC: Self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA of the hip and/or knee). The index consists of 24 questions (5 pain, 2 stiffness, and 17 physical function). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of to be replaced/replaced index joint (knee or hip) during past 48 hours. The WOMAC pain subscale score for each question ranges from 0 (minimum) to 4 (maximum), higher scores signifies worse pain. Pain subscale total score ranges from 0 to 20, with higher scores indicating worse pain.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Change From Baseline in Western Ontario and McMaster (WOMAC) Osteoarthritis Index Physical Function Subscale Score at Week 12
Description: WOMAC: Self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA of the hip and/or knee). Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in in the study joint during past 48 hours. The WOMAC physical function subscale score for each question ranges from 0 (minimum) to 4 (maximum), higher scores signifies worse physical function. Physical function subscale scores range from 0 to 68, where higher scores indicated more difficulty in performing daily activities.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Western Ontario and McMaster (WOMAC) Osteoarthritis Index Stiffness Subscale Score at Week 12
Description: WOMAC: Self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA of the hip and/or knee). Stiffness was defined as a sensation of decreased ease of movement in study joint. The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the in the study joint during the past 48 hours. The WOMAC stiffness subscale score for each question ranges from 0 (minimum) to 4 (maximum), higher scores signifies worse stiffness. The stiffness subscale score ranges from 0 to 8, where higher scores indicated worse stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Change From Baseline in Western Ontario and McMaster (WOMAC) Osteoarthritis Index Total Score at Week 12
Description: WOMAC: Self-administered, disease-specific questionnaire, which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA of the hip and/or knee). The WOMAC composite index was the sum of 24 individual questions regarding subscales of pain, stiffness and physical function (for each item score range: 0 [minimum] to 4 [maximum], higher score indicating worse study joint condition). Total score was sum of the 3 subscale scores, giving a possible overall score range of 0 (minimum) to 96 (maximum). Higher score indicating the worse level of pain, stiffness and physical function.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Change From Baseline in Knee Adduction Moment at Week 12
Description: Adduction (external) moment was defined as the ground-generated torque that forces the distal tibia toward the midline of the body, which forces the knee away from the midline, into a varus or "bow-legged" position. External knee adduction moment was assessed as percent body weight*height (%BW*ht).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Change From Baseline in Quadriceps Inhibition at Week 12
Description: Quadriceps inhibition was assessed in terms of flexion-extension range of motion and normalized mid stance knee flexion angle in degrees.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Change From Baseline in Peak Ground Reaction Force at Week 12
Description: Change from baseline in peak ground reaction force in body weight*seconds (BW*sec) was assessed with the help of a multicomponent force plate.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Change From Baseline in Total Ground Reaction Force at Week 12
Description: Change from baseline in total ground reaction force in body weight*seconds was assessed with the help of a multicomponent force plate.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Primary Outcome: Change From Baseline in Stride Length at Week 12
Description: The level walking was assessed by stride length; assessment was done based on 6 stride cycles over a range of walking speeds.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Primary Outcome: Change From Baseline in Walking Speed at Week 12
Description: Change from baseline in walking speed in meters per second was assessed.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Primary Outcome: Change From Baseline in Cadence at Week 12
Description: Cadence was defined as the rate at which a person walk, expressed in steps per minute.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: Change From Baseline in Patient Global Assessment of Arthritic Condition (PGAAC) Score at Week 12
Description: The PGAAC is self-administered measure in which participants answered the following question: "considering all the ways the OA in your signal knee affects you, how are you doing today?". Participants rated their condition using the following scale: 1= very good (no symptoms and no limitation of normal activities); 2= good (mild symptoms and no limitation of normal activities); 3= fair (moderate symptoms and limitation of some normal activities); 4= poor (severe symptoms and inability to carry out most normal activities); 5= very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated severe condition.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent to 28 days after the last study drug administration (up to 17 months)
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set population included all participants who received at least 1 dose of study medication.
Arm/Group | Placebo | Celecoxib 100 mg | Oxycodone 20 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Celecoxib 100 mg (N=6) | Oxycodone 20 mg (N=6)
Vision blurred (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Chills (General disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 3

LIMITATIONS AND CAVEATS:
No efficacy analysis were conducted, as this study was stopped due to a high screen failure rate before the planned enrollment required to carry out the pre-specified efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.